CLINICAL TRIAL: NCT06122220
Title: Optic Nerve Sheath Measurement and Angiogenic Factors for the Diagnosis of Pre-eclampsia
Brief Title: Optic Nerve Sheath Measurement and Angiogenic Factors in Patients With Pre-eclampsia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head of the research deparment, Saint Thomas Hospital, Panama
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FA012023
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pre-Eclampsia
Keywords: Angiogenic factors; Optic nerve sheath diameter; Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-eclampsia (Experimental): Subjects admitted with severe pre-eclampsia, based on the criteria by the American College of Obstetricians and Gynecologists (ACOG)
  Interventions: Procedure: ONSD+AF
- Control (Active Comparator): Subjects admitted for normal labor, without any criteria of pre-eclampsia
  Interventions: Procedure: ONSD+AF

INTERVENTIONS:
Procedure: ONSD+AF — Measurement of the optic nerve sheath diameter and of sFLT-1/PGIF index

SUMMARY:
Hypertensive disorders of pregnancy (HPT) are an important cause of maternal-feto-neonatal morbidity and mortality, being one of the three leading causes of maternal death in our country and in developing countries. The only cure for THE is termination of pregnancy, which ends up being a decision in which gestational age and maternal risks must be balanced. Angiogenic factors have come to occupy an indispensable place in the arsenal of tools that can be used to separate the patient with a high likelihood of complications from those in whom prolongation of pregnancy could represent an important neonatal benefit. Refining the diagnostic capability of this test would further improve maternal-fetal outcomes and the use of optic nerve sheath diameter (ONSD) measurement could make the difference.

The purpose of the present study is to correlate the measurement of ONSD with serum angiogenic factor (AF) values in patients with pre-eclampsia and to determine its predictive ability for adverse perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 24 and 40 weeks of gestation.

Exclusion Criteria:

* Multiple gestation
* Maternal vasculitis
* Previous cesarean section (3 or more)
* Brain or eye tumors
* Neurological conditions
* Chronic renal disease
* Purpura
* Heart disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter cut off value | Up to discharge. On average, 7 days.
  Value in mms of the optic nerve sheath diameter for the diagnosis of severe preeclampsia
sFLT-1/PiGF index | Up until discharge. On average, 7 days
  Value of the index between the sFlt-1/PIGF (angiogenic factor) for the diagnosis of severe preeclampsia

SECONDARY OUTCOMES:
Maternal/fetal morbidity | Up until discharge. On average, 7 days
  Presence of any/several indicators of maternal or fetal morbidity (abruptio placenta, HELLP syndrome, eclampsia, fetal growth restriction, acute lung edema).
Neonatal morbidity | Up until discharge. On average, 3 days
  Presence of any/several indicators of neonatal morbidity (Apgar scores, admission to NICU, encephalophatic hypoxia)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas Hospital, Panama City, Provincia de Panamá, Panama

IPD SHARING:
Plan to Share IPD: No